CLINICAL TRIAL: NCT05710068
Title: RF Microneedle Therapy Maintains the Treatment Effect of Melasma: A 32-week, Prospective, Randomized Split-face Study
Brief Title: Effects of RF Microneedle on Photoaging Skin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Jin Cheol Kim, Principal Investigator, Clinical Fellow, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AJOUIRB-INT-2021-133
Record Dates: First submitted 2023-01-13; First posted 2023-02-02 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Pigmentation; Pigmentation Disorder
MeSH Terms: conditions — Pigmentation Disorders | interventions — Lidocaine, Prilocaine Drug Combination

STUDY DESIGN:
Intervention Model Description: split lesion study
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional therapy with RF microneedle (Experimental): Half face Oral tranexamic acid combined with triple combination cream with RF microneedle
  Interventions: Device: RF Microneedle; Drug: Combination cream
- Conventional therapy (Active Comparator): Half face Oral tranexamic acid combined with triple combination cream
  Interventions: Drug: Combination cream

INTERVENTIONS:
Device: RF Microneedle — Pulsed-type RF device in bipolar mode with 25 non-insulated microneedles every 2 weeks for 6 month
  Arms: Conventional therapy with RF microneedle
Drug: Combination cream — 5% hydroquinone, 0.003% tretinoin, and 1% hydrocortisone twice daily for 2 months

SUMMARY:
Melasma relapse is almost common after discontinuation of conventional treatment. Recent studies have suggested that photoaging dermis is main pathomechanism of melasma emphasizing stromal targeting therapy. Therefore, we investigated maintenance effect of microneedle radiofrequency (RF) for melasma treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult more than 19 years old
* Melasma clinically diagnosed by three dermatologists

Exclusion Criteria:

* Aesthetic medical procedures in three months prior to the study
* Use of topical depigmenting agents in three months prior to the study
* Pregnant or lactating

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Change of modified melasma area severity index score | Every 1 month up to 8 months
  Change of modified melasma area severity index score
Change of lightness value | Every 1 month up to 8 months
  Change of lightness value by a chromometer

CONTACTS AND LOCATIONS:
Locations (1):
- Ajou University Hospital, Suwon, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Han HJ, Kim JC, Park YJ, Kang HY. Targeting the dermis for melasma maintenance treatment. Sci Rep. 2024 Jan 10;14(1):949. doi: 10.1038/s41598-023-51133-w. PMID 38200171